CLINICAL TRIAL: NCT04794127
Title: A Phase II Study on Trabectedin in Combination With PPARg Agonist Pioglitazone in Patients With Round Cell Myxoid Liposarcomas or Dedifferentiated G1 and G2 Liposarcomas With Stable Disease After a Monotherapy With Trabectedin. (TRABEPIO)
Brief Title: Study on Trabectedin in Combination With Pioglitazone in Patients Myxoid Liposarcomas With Stable Disease After T Alone.
Acronym: TRABEPIO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Humanitas Hospital, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-SARCO-7953
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-10

CONDITIONS: Liposarcoma, Myxoid; Liposarcoma, Dedifferentiated; Liposarcoma, Round Cell
Keywords: liposarcoma; trabectedin; pioglitazone
MeSH Terms: conditions — Liposarcoma, Myxoid; Liposarcoma | interventions — Trabectedin; Pioglitazone

STUDY DESIGN:
Intervention Model Description: Phase II, pilot, open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trabectedin in combination with Pioglitazone (Experimental): Trabectedin administered at a dose of 1.5 mg/m2-1.3 mg/m2 (according to investigator's choice, with a top-dose of 2.6 total mg per cycle) as a 24-hour continuous infusion via a central venous access every 3 weeks and Pioglitazone given continuously at the daily dose of 45 mg by oral route. Since Trabectedin has no cumulative toxicities, and Pioglitazone as well, the combination will be administered until progressive disease, major toxicity, patient's intolerance or unwillingness to continue treatment, or medical decision by the responsible physician.
  Interventions: Drug: Trabectedin; Drug: Pioglitazone Oral Product

INTERVENTIONS:
Drug: Trabectedin — Patients will be treated with Trabectedin administered at a dose of 1.5 mg/m2-1.3 mg/m2 (according to investigator's choice, with a top-dose of 2.6 total mg per cycle) as a 24-hour continuous infusion via a central venous access every 3 weeks and pioglitazone given continuously at the daily dose of 45 mg by oral route.
  Other Names: Trabectedine
Drug: Pioglitazone Oral Product — Patients will be treated with Trabectedin administered at a dose of 1.5 mg/m2-1.3 mg/m2 (according to investigator's choice, with a top-dose of 2.6 total mg per cycle) as a 24-hour continuous infusion via a central venous access every 3 weeks and pioglitazone given continuously at the daily dose of 45 mg by oral route.
  Other Names: Pioglitazone

SUMMARY:
This is a phase 2 study conducted in two sequential stages:

The first stage is an Italian single institution, single arm, pilot study, aimed at exploring the activity of the combination T and P in myxoid liposarcoma patients who achieved a stable disease after a minimum of 4 cycles of T alone. If a minimum required activity will be demonstrated from the first stage, the second stage of the study will be conducted;otherwise, the study will be stopped. The second stage is an Italian open-label, multicenter, randomized, double arm, phase II trial, aimed at evaluating the combination of T and P in myxoid liposarcoma and G1 or G2 dedifferentiated liposarcomas compared to the standard treatment with T alone. Patients will be randomized with a 1:1 ratio to treatments arms as specified below:

* Control arm (A): T alone
* Experimental arm (B): T in combination with P

DETAILED DESCRIPTION:
In the specific the first stage will be an Italian mono-institutional, single arm, pilot study exploring the activity of the combination of T and P in myxoid liposarcoma patients who achieved a stable disease after a minimum of 4 cycles of T alone. If a minimum required activity will be demonstrated from the first stage, the second stage of the study will be conducted; otherwise, the study will be stopped.

The second stage will be an Italian multicenter, open-label, randomized, double arm, phase II trial, aimed at evaluating the combination of T and P in myxoid liposarcoma and G1 or G2 dedifferentiated liposarcomas compared to the standard treatment. Patients will be randomized by a centralized computer system with a 1:1 ratio to one of the following two arms:

* Control arm (A): T alone
* Experimental arm (B): T in combination with P The pilot study will be conducted in Italy at Istituto Nazionale Tumori Milano in order to recruit 10 evaluable patients. The second stage will be conducted in approximately 10 italian centers in order to recruit 80 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of myxoid/round cell liposarcomas
2. Histological diagnosis confirmation by a reference centre
3. Age ≥ 18 years
4. ECOG PS ≤2
5. One or more previous systemic treatments employing anthracyclines +/- ifosfamide (unless one or both are clinically contraindicated)
6. Four or more previous cycles of T with a stable disease as defined by RECIST criteria
7. Recovery from toxic effects of prior therapies to NCI CTC Grade 1 or higher
8. Provision of signed informed consent

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. Partial response or progression disease as per RECIST criteria to the previous treatment with T
3. Inadequate haematological, renal and liver functions
4. History of other malignancies (except basal cell carcinoma or cervical carcinoma in situ, adequately treated), unless in remission from 5 years or more and judged of negligible potential of relapse
5. Known central nervous system (CNS) metastases
6. Active viral hepatitis or chronic liver disease
7. Unstable cardiac condition, including congestive heart failure or angina pectoris, myocardial infarction within one year before enrolment, uncontrolled arterial hypertension or arrhythmias
8. Active major infection
9. Other serious concomitant illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Objective response (OR) in patients with myxoid liposarcomas according to RECIST criteria or CHOI criteria | From the date of the enrollment up to 24 months
  The primary activity endpoint is the number of responders. Patients will be considered as responders if they reach a CR or PR as best response during treatment according to RECIST criteria or according to Choi criteria.

SECONDARY OUTCOMES:
Number and severity of Adverse Events | up to 24 months
  The safety profile of T+P is assessed by the frequency and type of treatment emergent adverse events, graded according to NCI-CTCAE v5.0, frequency and nature of SAEs.
Maximum Plasma Concentration [Cmax] | up to 24 months
  The analysis of [Cmax] will be performed on the first four enrolled patients within the safety analysis set 1.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio D'Incalci, MD, Study Chair — Humanitas University; Irene De Simone, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No